CLINICAL TRIAL: NCT02496494
Title: The Effects of Conversion From Cyclosporine to Tacrolimus on the Changes of Cardiovascular Risk Profiles and Serum Metabolites in Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Duck Kim, M.D., Ph.D., Associate Professor, Kyungpook National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNUH 2012-09-010
Record Dates: First submitted 2015-07-03; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: CYCLOSPORINE/TACROLIMUS
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus conversion group (Experimental): Cyclosprine was converted to tacrolimus in kidney transplant recipients.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus for maintenance immunosupression in kidney transplant recipients
  Other Names: TacroBell

SUMMARY:
The purpose of this study is to evaluate the effects of conversion from cyclosporine to tacrolimus on the changes of cardiovascular risk profiles and serum metabolites in renal transplant recipients.

DETAILED DESCRIPTION:
During the past two decades, cyclosporine has proved to be a valuable immunosuppressive drug that has contributed to a significant reduction in the incidence of acute rejection after kidney transplantation. However, cyclosporine is known as a major factor causing cardiovascular death in kidney transplant recipients. Moreover, cyclosporine has an adverse effect on the lipid profile and fibrinolytic system and result in hypertension and cardiovascular disease. Immunosupressive mechanism of tacrolimus is identical that of cyclosporine but it is 100 times more potent T cell inhibitor than cyclosporine. In multicenter study of Europe and United states, tacrolimus showed low incidence of acute rejection and was known to effective in acute rejection resistant to other therapy. Tacrolimus has a lot of advantages compared to cyclosporine in terms of hypertensive and hyperlipidemic effects although evidences are lacking. One study demonstrated cardiovascular risk profile and renal function has been improved in kidney transplant patients after randomized conversion from cyclosporine to tacrolimus Previous study analyzing metabolites of tacrolimus and cyclosporine revealed that differences were observed in the metabolite level of hypoxanthine, lactate, succinate, and taurine between two immunosupressants. The objective of this study is to evaluate changes in cardiovascular risk profiles and metabolite patterns after conversion from cyclosporine to tacrolimus in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received a kidney transplant at least 12 months ago prior to enrollment
2. Patients who have kept in unchanged cyclosporine therapy at least for 6 months prior to enrollment.
3. Female patients of childbearing potential must have a negative urine or serum pregnancy test prior to enrollment, and agreed to the deliberate prevention of conception during the trial
4. Patients who are considered clinically stable by observer's judgment.
5. Patients must understand the purpose and risk of participating the the trial and signed on the written consent.

Exclusion Criteria:

1. Patients who have previously received an organ transplant other than a kidney
2. Patients diagnosed with congestive heart failure within 6 months (EF <35%)
3. Patients with untreated ischemic heart disease
4. Patients whose hemoglobin is in the level of <7.0 g/dL
5. Patients who have a known hypersensitivity to tacrolimus
6. Patients taking potassium sparing diuretics
7. Patients newly diagnosed malignant tumors after organ transplant but the patients treated completely with basal or squamous cell carcinoma of the skin are excepted
8. Patients who are at the risk of drug abuse or mental disorders or communicate difficulties with the observer
9. Patients who are pregnant or lactating

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Blood Pressure at 6 months | 3 months, 6 months
Change from Baseline in Lipid Profile at 6 months | 3 months, 6 months

SECONDARY OUTCOMES:
Assessing glucose regulation using blood glucose and hemoglobin A1c | 3 months, 6 months
Assessing other metabolic cardiovascular risk factors using fibrinogen, tPA, PAI-I, homocysteine, pro-BNP, hs-CRP, uric acid | 24 weeks
Assessing serum metabolite using ELISA | 3 months, 6 months
Assessing renal function using blood urea nitrogen and creatinine | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Duck Kim, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea